CLINICAL TRIAL: NCT06309758
Title: BreinZorg: A Feasibility Study Into an Online Lifestyle Platform for Mild Cognitive Impairment (MCI) and Subjective Cognitive Decline (SCD)
Brief Title: BreinZorg: Feasibility Study Into an Online Lifestyle Platform for MCI and SCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 115022
Record Dates: First submitted 2024-02-21; First posted 2024-03-13 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-01

CONDITIONS: Mild Cognitive Impairment; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: mixed-method study with a single-arm pre-post design with a duration of 3 months and extended follow-up after 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): 3 month active use of the website. Receive bi-weekly update mails to nudge participants to use the website.
  Interventions: Other: Breinzorg

INTERVENTIONS:
Other: Breinzorg — The BreinZorg multidomain lifestyle website comprises 16 domains, namely (1) physical activity, (2) healthy diet, (3) smoking, (4) alcohol, (5) sleep, (6) cognitive activity (7) social activity, (8) diabetes, (9) blood pressure, (10) cholesterol, (11) heart- and vascular diseases, (12) kidney diseases, (13) hearing damage, (14) obesity, (15) anxiety, and (16) depression. These 16 modules are separated into three big themes: mood, lifestyle, and body.
  Each module consists of the following:
  1. General information on the risk factor;
  2. Tips on how to improve and decrease the risk;
  3. Quiz questions about the risk factor, giving extra knowledge/ in a playful and interactive manner;
  4. Examples of SMART goals fitting the risk factor (goal examples are given in a Specific, Measurable, Achievable, Relevant, and Time-Bound manner).

SUMMARY:
Dementia is the most common disease in older individuals and this century's biggest healthcare challenge. Many patients who visit the memory clinic with memory complaints do not have dementia but instead are diagnosed with mild cognitive impairment (MCI) or subjective cognitive decline (SCD). MCI or SCD may be a pre-dementia stage. Many patients with MCI or SCD often leave their consultation with unanswered questions, and unsure what they, themselves can do to reduce dementia risk. Patients with MCI and SCD have a heightened risk of developing dementia. Therefore, this group would possibly benefit most from preventive strategies. Around 40% of dementia cases is attributable to modifiable factors. Thus, managing a healthy lifestyle may reduce dementia risk.

To answer the information request many patients have when leaving the memory clinic and to fill the knowledge gap an online tool has been developed.

The goal of this mixed-method feasibility study is to investigate the usability, feasibility, patient experience, and effectiveness of the personalized, multi-domain online website in older adults with MCI or SCD.

The main questions it aims to answer are:

* Is the new website being used by the target population?
* How does the target population experience the use of the website?
* What is the effect of using the website?

Participants will have access to the website and are free to use the website in any way they want.

ELIGIBILITY:
Inclusion Criteria:

* Visited a memory clinic;
* Recent (no longer than 4 months) diagnosis of MCI or SCD according to the guidelines used in the memory clinic;
* >60 years of age;
* Sufficient fluency in Dutch;
* Internet access at home and a working e-mail address;
* Sufficient hearing and vision to read, watch and hear content on the website.

Exclusion Criteria:

* Diagnosis of Dementia according to the guidelines of the memory clinic;
* Any condition to hinder successful 6-month follow-up;
* Diagnosis of Major depression;
* Coincident participation in any other intervention trial at time of pre-screening.

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the new online website following the theoretical framework of acceptability | After 3 months
  The perception among the patients that the intervention (website) is agreeable. The investigators collect data by means of a questionnaire following the theoretical framework of acceptability. Assessing 7 constructs of acceptability: Affective attitude, Burden, Ethicality, Perceived effectiveness, intervention coherence, self-efficacy and, opportunity costs. Additionally, qualitative information is on experiences and acceptability is gathered using semi-structured interviews.
Adoption / Uptake of the new online website. Website usage data. | After 3 months and after 6 months
  The intention, initial decision, or action to try to employ a new intervention. How much and how is the new website used by the participants? The investigators collect monitoring data of the website on usage of the website.
Demand of the new online website. Website usage data. | After 3 months and after 6 months
  The estimated use or actual use of the intervention.Monitoring data on the use of the website. How much time do participants spend on the website, which pages do they use and how many times do they visit the website?
Practicality of the new online website. | After 3 months
  The extent to which the intervention can be delivered. Interviews in a subgroup will contain questions on the burden and barriers of the website. It will also contain questions on the desired frequency, duration, and intensity of the website.
Feeling of trust in yourself and your own abilities. | At baseline, after 3 months and after 6 months
  Effectiveness of the website in increasing feelings of self-efficacy. This is measured by the General Self-Efficacy Scale (GSES) questionnaire.
  The scale goes from 'totally do not agree' to 'totally agree'. A higher score on this questionnaire means the participant has more feeling of trust in themselves and their abilities. scores will range between 10 and 50.
Feeling of control about own life and future. | At baseline, after 3 months and after 6 months
  Effectiveness of the website in increasing feeling of control. This is measured by the 7-item Pearlin Mastery Scale.
  The scale goes from 'totally do not agree' to 'totally agree'. A higher score on this questionnaire means the participant has more feeling of control. scores will range between 7 and 35.
Motivation to change lifestyle for reduction of dementia risk. | At baseline, after 3 months and after 6 months
  Effectiveness of the website in increasing motivation to make lifestyle changes. This is measured by the Dutch Motivation to Change Lifestyle and Health Behaviours for Dementia Risk Reduction (MCLHB-DRR) questionnaire.
  The answers to this questionnaire will result in 8 different scores. A score for perceived susceptability, perceived severity, perceived barrieres, perceived benefits, cues to action, general health motivation, self-efficacy, and a total motivation.
  A higher score means more motivation. The scale goes from 'totally do not agree' to 'totally agree'. scores will range between 27 and 135.
Awareness about dementia risk reduction | At baseline, after 3 months and after 6 months
  effectiveness of the website in increasing awareness and knowledge on dementia risk reduction. This is measured by a modified version of the awareness survey that has been used in the 'MijnBreinCoach' study. This questionnaire focuses on knowledge about dementia risk reduction by changing lifestyle factors.
  A higher score means more awareness and knowledge on dementia risk reduction. The scale goes from 'totally do not agree' to 'totally agree'. scores will range between 16 and 80.

SECONDARY OUTCOMES:
Change in alcohol consumption | At baseline, after 3 months and after 6 months
  The efficacy of the website in changing a user's consumption of alcohol. This is measured by our questionnaire asking about the consumption of the participant. The change in answers will be an indication that website is successful in changing alcohol consumption.
Change in smoking behaviour | At baseline, after 3 months and after 6 months
  The efficacy of the website in changing a user's smoking behavior. This is measured by our questionnaire asking about the smoking behavior of the participant. The change in answers will be an indication that the website is successful in changing smoking behavior.
Change in physical exercise. | At baseline, after 3 months and after 6 months
  physical activity of a participant is assessed with the Short Questionnaire to Assess Health-enhancing Physical Activity (SQUASH). The change in scores/answers will be an indication that the website is effective in changing someone's physical activity.
Change in Diet. | At baseline,after 3 months and after 6 months
  Diet will be assessed with the Mediterranean Diet Adherence Screener (MEDAS). This will assess if the participant follows a Mediterranean diet or not. The change in the score on the MEDAS will indicate if a participant has changed their diet to be more like a Mediterranean diet. This will be an indication that the website is effective in changing a participant's diet.
  Scores on the MEDAS questionnaire will range between 0 and 14. A higher score means that the participants follows the mediterranean diet more closely.
Change in Sleep behaviour | At baseline, after 3 months and after 6 months
  Sleep behavior will be assessed by means of the Pitsburg Sleep Quality Index (PSQI). The change in answers on the PSQI will indicate if a participant's sleep pattern and behavior have changed. This will be an indication that the website is effective in changing a participant's sleep behavior.
Change in cognitive activities. | At baseline, after 3 months and after 6 months
  A participant's cognitive activities are assessed with the Cognitive and Leisure Activity Scale (CLAS). A change in this score will indicate if a participant has taken on more or less cognitive activities after using the website. This will be an indication that the website is effective in changing the amount of cognitive activities a participant undertakes.
  Answers on the CLAS go from 'never' to 'daily' and the scores will range between 11 and 66. A higher score on the CLAS indicates more cognitive activities for the participants.
Change in Stress levels | At baseline, after 3 months and after 6 months
  Stress is assessed by the Perceived Stress Scale (PSS). A change in scores on the PSS will indicate if a participant feels more or less stressed. This may be an indication that our website is effective in changing the amount of stress a participant feels.
  Answers to the PSS questions range from 'never' to 'really often (zeer vaak in dutch)'. The score will range from 10 to 50 and a higher score means the participants has less stress.
Change in Mental health Quality of Life | At baseline, after 3 months and after 6 months
  Quality of life will be assessed using the Mental Health Quality of Life (MHQoL) questionnaire. This questionnaire focuses more on the mental health aspect of quality of life, such as mood, self-image, and feelings toward the future. A change in this score indicates a feeling of a better or worse Quality of life. This may also indicate that our website is effective in changing this feeling.
  Questions on the MHQoL have all different answers, they ask about different things such as relations, health and future. The answers are an indication how the participants feels. The score will range between 8 and 32, where a higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
plan to share, but no IPD sharing plan ready.